CLINICAL TRIAL: NCT04847830
Title: Effects of Adjunctive Er, Cr :YSGG Laser Treatment to Nonsurgical Periodontal Treatment on Healing of Intrabony Periodontal Defects: a Randomised Controlled Trial
Brief Title: Adjunctive Laser for Periodontal Intrabony Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 276918
Record Dates: First submitted 2021-04-01; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Lasers, Solid-State

STUDY DESIGN:
Intervention Model Description: non-surgical periodontal therapy with or without laser adjunct
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomisation for the site receiving the additional test procedure (laser) will be carried out between baseline and visit 2. The randomisation will be carried out by Postgraduate Students independent of the study. Random permuted block sizes of 4 will be employed. The centralised randomisation service 'Sealed envelope' will be used for randomisation and to ensure allocation concealment. A sealed envelope will be enclosed with the patient's notes by personnel not directly involved in the study. The therapist will only be informed about treatment allocation by opening the envelope following completion of non-surgical therapy (when the laser will need to be employed on the test site). No minimization or stratification is planned. The randomisation code will only be revealed after statistical analysis. The randomisation will be done by a different postgraduate student who will be masked and is not involved in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser (Experimental): One side of the mouth will undergo root surface debridement using hand instruments and ultrasonic scaler, with the addition of the Er:YAG laser
  Interventions: Device: Er:YAG laser (Waterlase); Procedure: root surface dbridement
- Control (Placebo Comparator): The other side of the mouth undergo root surface debridement using hand instruments and ultrasonic scaler alone
  Interventions: Procedure: root surface dbridement

INTERVENTIONS:
Device: Er:YAG laser (Waterlase) — The WaterLase iPlus tissue cutting system is a unique device with diverse, hard- and soft-tissue dental applications. It utilizes advanced laser and water atomization technologies to safely and effectively cut, shave, contour, roughen, etch, and resect oral hard-tissue, and direct laser energy to perform oral soft-tissue removal, incision, excision, ablation and coagulation.
  Arms: Laser
Procedure: root surface dbridement — root surface debridement under local anaesthesia

SUMMARY:
Participants with periodontitis and presence of bilateral intrabony defect will be randomised to have one side of the mouth undergo root surface debridement using hand instruments and ultrasonic scaler alone, while the contralateral side will receive the same treatment, with the addition of the Er:YAG laser. Outcomes studies will be periodontal clinical parameters at 3 months, 6 months, 9 months and 12 months after treatment, radiographic parameters at 12 months, patient-reported parameters and laboratory analyses.

DETAILED DESCRIPTION:
The study is a Double-masked randomised controlled trial with split-mouth design.

Participants with periodontitis will be randomised to have one side of the mouth undergo root surface debridement using hand instruments and ultrasonic scaler alone, while the contralateral side will receive the same treatment, with the addition of the Er:YAG laser. Outcomes studies will be periodontal clinical parameters at 3 months, 6 months, 9 months and 12 months after treatment, radiographic parameters at 12 months, patient-reported parameters and laboratory analyses.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of 20 teeth. Diagnosis of Severe Periodontitis (Diagnosis of Periodontitis stage III or IV (grade A, B or C) (Tonetti et al. 2018)

Presence of at least 2 teeth with ≥ 6 mm pockets and minimum of 3 mm intrabony defect, in opposing quadrants of the upper or lower arch.

Exclusion Criteria:

* Inclusion:

Minimum of 20 teeth. Diagnosis of Severe Periodontitis (Diagnosis of Periodontitis stage III or IV (grade A, B or C) (Tonetti et al. 2018)

Presence of at least 2 teeth with ≥ 6 mm pockets and minimum of 3 mm intrabony defect, in opposing quadrants of the upper or lower arch.

Exclusion:

* Wearing of a removable appliance/denture
* Wearing of orthodontic appliances.
* Current smoking - any history of smoking or vaping within last 5 years
* Relevant medical history likely to affect periodontal disease or taking relevant medication, including diabetes, as judged by the examining clinician
* Periodontal treatment (surgical/non-surgical root surface debridement under local anaesthesia) within last 12 months, as judged by the examining clinician
* History of any antibiotic use within last 3 months.
* Pregnant patients
* Teeth with hopeless prognosis indicated for extraction (Cortellini et al 2011)
* Patients with a non-adequate level of English

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Pocket resolution | 12 months
  Number of sites with absence of PPD >5mm following adjunctive laser treatment with RSD (= no need for surgery)

SECONDARY OUTCOMES:
Gain bone height | 12 months
  Radiographic improvement in bone levels
Patient-related outcomes | 12 months
  Questionnaire-based patient-reported outcomes
GCF biomarkers | 12 months
  Change in GCF concentration Biomarkers
Recession | 12 months
  Changes in gingival recession measurement
CAL | 12 months
  Changes in clinical attachment level
Mobility | 12 months
  Changes in mobility scores

IPD SHARING:
Plan to Share IPD: No